CLINICAL TRIAL: NCT01686893
Title: STIT-1 Evaluation of Safety and Efficacy of Shorttime TNI Treatment in Patients With COPD
Brief Title: Evaluation of Safety and Efficacy of Shorttime TNI Treatment in Patients With COPD
Acronym: STIT-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Christian M. Kaehler, Head of Pneumology, Clinical Professor, Medical University Innsbruck
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AN3547; AN 3546 (Other: Ethics Committee Innsbruck)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Oxygen Inhalation Therapy
Keywords: Oxygen, Insufflation, COPD, High Flow Treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Nasal Insufflation of oxygen (Active Comparator): Standard Nasal Insufflation of oxygen
  Interventions: Device: Standard Nasal Insufflation of oxygen
- Nasal oxygen insufflation with a TNI 20 oxy device (Active Comparator): Nasal oxygen insufflation with a TNI 20 oxy device
  Interventions: Device: Nasal oxygen insufflation with a TNI 20 oxy device

INTERVENTIONS:
Device: Nasal oxygen insufflation with a TNI 20 oxy device — Nasal oxygen insufflation with a TNI 20 oxy device
  Other Names: TNI 20 oxy
  Arms: Nasal oxygen insufflation with a TNI 20 oxy device
Device: Standard Nasal Insufflation of oxygen — Standard Nasal Insufflation of oxygen
  Arms: Standard Nasal Insufflation of oxygen

SUMMARY:
Evaluation of Safety and Efficacy of Shorttime TNI Treatment in Patients with COPD Acute testing of oxygen demand using TNI vs. standard oxygen application in stable COPD patients An investigator-initiated, prospective, controlled, multicenter study

DETAILED DESCRIPTION:
TNI, the nasal insufflation of a high flow of warm, humidified air, is an extremely comfortable and uncomplicated alternative to numerous other approaches in non-invasive ventilation (NIV). Up to now, NIV therapy could only be applied by masks with the associated complications as patients could not tolerate high airflow delivered by a thin nasal cannula without humidification and warming, thus causing concomitant negative effects. The new therapy TNI shows a high rate of acceptance by children, too.

At present, there are two different types of devices available for nasal insufflation in clinics:

TNI 20s, an air humidifier for clinical compressed air, and the TNI20 oxy, an air humidifier for clinical compressed air, which can be combined with oxygen.

TNI 20 oxy The system, which is unique throughout the world, is optimized for the application of flows of up to 20L/min and fulfils the minimum requirements of the "American Society of Testing and Materials" for a high flow air humidifier in the non-invasive application of 10 mg H2O/L (equivalent to about 60% rel. humidity at an ambient temperature of 22°C) for the air humidity. The warming of the air flow by 5-15°C can be adjusted relative to the ambient temperature. Condensation is prevented in the nasal applicator by heating the tube as far as the nostrils. The device automatically controls humidity and temperature depending on the prevailing ambient conditions. The TNI®20s can be attached to the hospital infrastructure by means of a standard pressure regulator.

ELIGIBILITY:
Inclusion Criteria:

- COPD patients with an indication for long-term oxygen therapy Age 30 - 80 years COPD GOLD °III

Exclusion Criteria:

- Clinical instability of the patient No lung function testing possible Exacerbation within the last 14 days prior to inclusion into the study Serious concomitant diseases that may jeopardize the inclusion of the patient into the study from the investigator's point of view Anaemia, defined by a haemoglobin <10 G/L Patients with hypercapnia, defined by a paCO <46mmHg Participation of the patient in any other ongoing study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
PaO2 | Measures at Baseline and after 60 min
  Change in the partial oxygen pressure in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)

SECONDARY OUTCOMES:
O2 % | Measures at Baseline and after 60 min
  Change in the oxygen saturation in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)
PaCO2 | Measures at Baseline and after 60 min
  Change in the partial carbon dioxide pressure in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)
AaDO2 | Measures at Baseline and after 60 min
  Change in the AaDO2 in the peripheral blood at a defined oxygen flow rate (L/min)
RV and TLC | Measures at Baseline and after 60 min
  Safety of the device in COPD °III or IV patients:
  No increase in the residual volume (RV) and the total lung capacity (TLC) > 15% of the mean actual value at visits 1 and 2 (measurement 60 + 10 minutes after oxygen insufflation with a TNI system).

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Kaehler, MD, Principal Investigator — Pneumology, Medical University Innsbruck
Locations (3):
- Pneumology/USPH Innsbruck, Medical University Innsbruck, Innsbruck, Austria
- Pneumologie, Medizinische Klinik und Poliklinik I, University Dresden, Dresden, Germany
- Klinik und Poliklinik für Pneumologie, Inselspital, Universitätsspital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Vogelsinger H, Halank M, Braun S, Wilkens H, Geiser T, Ott S, Stucki A, Kaehler CM. Efficacy and safety of nasal high-flow oxygen in COPD patients. BMC Pulm Med. 2017 Nov 17;17(1):143. doi: 10.1186/s12890-017-0486-3. PMID 29149867